CLINICAL TRIAL: NCT05425784
Title: Regular Home Use of Dual-light Photodynamic Therapy in the Management of Chronic Periodontitis
Brief Title: Home Use of Dual-light Photodynamic Therapy for Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koite Health Oy (Industry)
Collaborators: University of Helsinki (Other); University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LumoNorth2022
Record Dates: First submitted 2022-05-31; First posted 2022-06-21 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Periodontal Diseases; Periodontitis; Plaque, Dental; Plaque Induced Gingivitis
Keywords: Lumoral; Lumorinse; Plaque; Periodontitis; Plaque control; aPDT; aMMP-8
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Dental Plaque; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: 90 participants are randomized into two arms: the Lumoral-treatment arm and Control arm.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The subjects will be randomized to the study group and the control group by using a sealed envelope system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumoral Treatment (Study group) (Experimental): Subjects will receive detailed instructions for the use of Lumoral treatment -device and Lumorinse -tablets. Subjects will be instructed to use the Lumoral treatment -device and follow the protocol five to seven (5-7) times a week. Regular use shall be defined as frequency of a minimum of twice a week.
  Standard oral hygiene instructions will be provided verbally and in writing. In addition, an electric toothbrush will be provided to all subjects.
  Interventions: Device: Lumoral treatment; Other: Standard oral hygiene self care
- Standard of care (Control group) (Active Comparator): Standard oral hygiene instructions will be provided verbally and in writing. In addition, an electric toothbrush will be provided to all subjects.
  Interventions: Other: Standard oral hygiene self care

INTERVENTIONS:
Device: Lumoral treatment — The investigational Lumoral treatment -device provides a constant and repeatable application which can be done at home and is easily available. All subjects in the study group will receive their own Lumoral treatment -device and Lumorinse-mouth rinse tablets for the complete duration of the study.
  Other Names: Lumorinse mouth rinse
  Arms: Lumoral Treatment (Study group)
Other: Standard oral hygiene self care — Both groups shall be given oral and written instructions for twice-daily standard oral hygiene self-care.
  Other Names: Electric toothbrush provided

SUMMARY:
This early-stage research is designed to determine the efficacy of the Lumoral method in chronic periodontitis patients. Improved supragingival plaque control can help to also sustain the subgingival plaque management in the long term. In addition, the device might have a photobiomodulation effect on periodontal tissues.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease leading to a progressive loss of the tooth-supporting apparatus. The disease is strongly associated with deranged biodiversity patterns in dental plaque.

The Lumoral is a CE-marked medical device developed to provide a potent, targeted antibacterial action on dental plaque in a home environment. The device mechanism of action is antibacterial photodynamic therapy. The device is used by swishing a mouth rinse, which has a strong adherence to dental plaque. The plaque-adhered photoactive mouth rinse can be activated by a simple to use light applicator. The antibacterial efficacy far exceeds chlorhexidine, without side effects in a longterm use. Preliminary results have shown a promising anti-inflammatory response in addition to plaque reduction.

Ninety (90) stage I-III periodontitis patients are randomized to Lumoral treatment group or control group. Both groups shall receive mechanical plaque control by scaling and root planning (SRP) and standard oral hygiene instructions for electric toothbrush, interdental brush, and dental floss use. All the patients shall be assessed for the clinical periodontitis status. These assessment and analyses shall be performed at baseline, at 3 months and at 6 months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal disease stage I-III, according to criteria the American Academy of Periodontology (AAP) with at least 2 mm interdental CAL in the site of greatest loss.
* Age of 18- 85 years
* Presence of ≥20 teeth, including implants
* Agreement to participate in the study and to sign a written consent form
* Able to co-operate with the treatment protocol and avoid any other oral hygiene measures outside of the study protocol

Exclusion Criteria:

* Presence of major physical limitation or restriction that prohibit the hygiene procedures used in the study protocol
* Removable major prosthesis or major orthodontic appliance
* Pregnancy or lactation
* Use of antibiotics within 2 weeks prior the study
* A need for immediate antimicrobial treatment for periodontitis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Reduction in dental inflammation | 3 months
  Possible changes in dental inflammation measured by bleeding on probing (BoP) when compared to control group at 3 months compared to baseline
Reduction in dental inflammation | 6 months
  Possible changes in dental inflammation measured by bleeding on probing (BoP) when compared to control group at 6 months compared to baseline
Stabilization of the periodontal disease | 3 months
  Possible changes in the periodontal disease, measured by total probing pocket depth (PPD) progression in the patient mouth at 3 months compared to baseline
Stabilization of the periodontal disease | 6 months
  Possible changes in the periodontal disease, measured by total probing pocket depth (PPD) progression in the patient mouth at 6 months compared to baseline

SECONDARY OUTCOMES:
Reduction in aMMP-8 measurement | 3 months
  Clinical improvement in periodontal inflammation marker aMMP-8 measured by Periosafe® at 3 months compared to baseline
Reduction in aMMP-8 measurement | 6 months
  Clinical improvement in periodontal inflammation marker aMMP-8 measured by Periosafe® at 6 months compared to baseline
Improvement in probing pocket depth (PPD) reflecting the clinical periodontitis status | 3 months
  Clinical improvement of periodontitis measured by probing pocket depth (PPD) at 3 months based on the absolute values of PPD. All clinical parameters will be recorded with the help of a graded periodontal manual probe (for example, North Carolina 54B or UNC15 probe (Hu-Friedy Mfg. Co., LLC) or similar device) with a maximum force of 0.25 N.
Improvement in probing pocket depth (PPD) reflecting the clinical periodontitis status | 6 months
  Clinical improvement of periodontitis measured by probing pocket depth (PPD) at 6 months based on the absolute values of PPD. All clinical parameters will be recorded with the help of a graded periodontal manual probe (for example, North Carolina 54B or UNC15 probe (Hu-Friedy Mfg. Co., LLC) or similar device) with a maximum force of 0.25 N.
Improvement in clinical attachment level (CAL) reflecting the clinical periodontitis status | 3 months
  Clinical improvement of periodontitis measured by clinical attachment level (CAL) at 3 months based on the absolute values of CAL. All clinical parameters will be recorded with the help of a graded periodontal manual probe (for example, North Carolina 54B or UNC15 probe (Hu-Friedy Mfg. Co., LLC) or similar device) with a maximum force of 0.25 N.
Improvement in clinical attachment level (CAL) reflecting the clinical periodontitis status | 6 months
  Clinical improvement of periodontitis measured by clinical attachment level (CAL) at 6 months based on the absolute values of CAL. All clinical parameters will be recorded with the help of a graded periodontal manual probe (for example, North Carolina 54B or UNC15 probe (Hu-Friedy Mfg. Co., LLC) or similar device) with a maximum force of 0.25 N.
Change in periodontal microbiological pathogens. | 3 months
  Clinical improvement in periodontal microbiological pathogens at 3 months compared to baseline. The microbiological evaluation is the Quantification of periodontopathic bacteria by 16S rRNA sequencing analysis. Microbiological sample will be collected using so called Iso Taper Paper Points, size-20 (VDW GmbH) from selected gingival/periodontal pockets with maximum initial probing depth. The paper points will then be be placed into sterile, small-aliquot containers, and immediately stored at -20°C until analysis.
Change in periodontal microbiological pathogens. | 6 months
  Clinical improvement in periodontal microbiological pathogens at 6 months compared to baseline. The microbiological evaluation is the Quantification of periodontopathic bacteria by 16S rRNA sequencing analysis. Microbiological sample will be collected using so called Iso Taper Paper Points, size-20 (VDW GmbH) from selected gingival/periodontal pockets with maximum initial probing depth. The paper points will then be be placed into sterile, small-aliquot containers, and immediately stored at -20°C until analysis.
Improvement in oral-related quality of life. | 3 months
  Patient related objectives: Improvement in oral-related quality of life measurement (OHIP-14) questionnaire at baseline, at 3 months compared to baseline.
  Fourteen items of OHIP are divided into seven dimensions: functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability, and handicaps. Grading is based on answering a five-scale questionnaire from 'Never' to 'Very often'.
Improvement in oral-related quality of life. | 6 months
  Patient related objectives: Improvement in oral-related quality of life measurement (OHIP-14) questionnaire at baseline, at 6 months compared to baseline.
  Fourteen items of OHIP are divided into seven dimensions: functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability, and handicaps. Grading is based on answering a five-scale questionnaire from 'Never' to 'Very often'.

CONTACTS AND LOCATIONS:
Overall Officials: Tommi Pätilä, Docent, Study Director — Chief Medical Officer; Timo Sorsa, Professor, Principal Investigator — University of Helsinki
Locations (3):
- Finland (3):
  - Mehiläinen Länsi-Pohja Central Hospital, Kemi, Lapland
  - Hammas Hohde Oy, Oulu, Oulun Lääni
  - City of Rovaniemi Health Cervices, Oral Health, Rovaniemi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alaijah, F., Morsi, A., Nasher, R. et al. Photobiomodulation therapy in the treatment of periodontal disease: a literature review. — https://link.springer.com/article/10.1007/s41547-019-00056-9
- See also: Joshi K, Baiju CS, Khashu H, Bansal S (2020) Clinical effectiveness of indocyanine green mediated antimicrobial photodynamic therapy as an adjunct to scaling root planing in treatment of chronic periodontitis- A randomized controlled clinical trial. — https://pubmed.ncbi.nlm.nih.gov/31783161/
- See also: Kassebaum NJ, Bernabé E, Dahiya M et al., (2014) Global burden of severe periodontitis in 1990- 2010: a systematic review and meta-regression. — https://pubmed.ncbi.nlm.nih.gov/25261053/
- See also: Kassebaum NJ, Smith AGC, Bernabé E, et al., (2017) Global, Regional and National Prevalence, Incidence, and Disability-Adjusted Life Years for Oral Conditions for 195 Countries, 1990-2015: A Systematic Analysis for the Global Burden of Diseases, Injuries — https://pubmed.ncbi.nlm.nih.gov/28792274/
- See also: Lang NP, Suvan JE, Tonetti MS (2015) Risk factor assessment tools for the prevention of periodontitis progression a systematic review. — https://pubmed.ncbi.nlm.nih.gov/25496279/
- See also: Levine JI. Medications that increase photosensititivity. FDA document Dec 1990. — https://www.fda.gov/media/75892/download
- See also: Loos BG & Needleman I (2020) Endpoints of active periodontal therapy. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7670400/
- See also: Monzavi A, Chinipardaz Z, Mousavi M, et al., (2016) Antimicrobial photodynamic therapy using diode laser activated indocyanine green as an adjunct in the treatment of chronic periodontitis: A randomized clinical trial. — https://pubmed.ncbi.nlm.nih.gov/26921460/
- See also: Nikinmaa S, Alapulli H, Auvinen P, et al. (2020) Dual-light photodynamic therapy administered daily provides a sustained antibacterial effect on biofilm and prevents Streptococcus mutans adaptation. — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0232775
- See also: Pereira PAB, Aho VTE, Paulin L, et al., (2017) Oral and nasal microbiota in Parkinson's disease. — https://pubmed.ncbi.nlm.nih.gov/28259623/
- See also: Sanz M, Herrera D, Kebschull M, et al.; On behalf of the EFP Workshop Participants and Methodological Consultants. (2020) Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline. — https://pubmed.ncbi.nlm.nih.gov/32383274/
- See also: Schär D, Ramseier CA, Eick S, et al., (2020) Transgingival photodynamic therapy (tg-aPDT) adjunctive to subgingival mechanical instrumentation in supportive periodontal therapy. A randomized controlled clinical study. — https://doi.org/10.1016/j.pdpdt.2020.101971
- See also: Slade GD (1997) Derivation and validation of a short-form oral health impact profile — https://pubmed.ncbi.nlm.nih.gov/9332805/